CLINICAL TRIAL: NCT05814939
Title: A Multicenter, Randomized, Double-blind, Controlled Phase II Clinical Study to Evaluate the Efficacy and Safety of VC005 Tablets in Subjects With Active Ankylosing Spondylitis.
Brief Title: Efficacy and Safety Clinical Study of VC005 Tablets in Subjects With Active Ankylosing Spondylitis.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jiangsu vcare pharmaceutical technology co., LTD (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: VC005-201
Record Dates: First submitted 2023-04-04; First posted 2023-04-18 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Active Ankylosing Spondylitis
MeSH Terms: interventions — tofacitinib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- VC005 Tablets Low Dose groups (Experimental)
  Interventions: Drug: VC005 tablets
- VC005 Tablets Medium Dose groups (Experimental)
  Interventions: Drug: VC005 tablets
- VC005 Tablets High Dose groups (Experimental)
  Interventions: Drug: VC005 tablets
- Tofacitinib Citrate Tablets groups (Active Comparator)
  Interventions: Drug: Tofacitinib Citrate Tablets
- VC005 Tablets Placebo groups (Placebo Comparator)
  Interventions: Drug: VC005 Tablets Placebo

INTERVENTIONS:
Drug: VC005 tablets — VC005 groups repeat administration for 12 weeks
  Arms: VC005 Tablets High Dose groups; VC005 Tablets Low Dose groups; VC005 Tablets Medium Dose groups
Drug: Tofacitinib Citrate Tablets — Tofacitinib Citrate groups repeat administration for 12 weeks
  Arms: Tofacitinib Citrate Tablets groups
Drug: VC005 Tablets Placebo — VC005 placebo groups repeat administration for 12 weeks
  Arms: VC005 Tablets Placebo groups

SUMMARY:
This clinical trial is a multicenter, randomized, double-blind, controlled phase II clinical study.

ELIGIBILITY:
Inclusion Criteria:

1. The subject understands and voluntarily signs the informed consent form (ICF) and is willing and able to comply with the study protocol;
2. The subject is between 18 and 70 years of age (including borderline values) at the time of signing the ICF, regardless of gender;
3. The subject has been diagnosed with AS according to the 1984 New York Revised Criteria for Ankylosing Spondylitis (AS can be diagnosed by having Article ④ and any one of Articles ① to ③): ① lower back pain lasting for at least 3 months, with pain improving with activity but not with rest; ② limited movement of the lumbar spine in the anterior-posterior and lateral flexion directions; ③ thoracic extension less than normal for the same age and sex; ④ bilateral sacroiliac arthritis grade II-IV, or unilateral sacroiliac arthritis grade III-IV;
4. The subject had active disease prior to the screening visit and randomization, defined as follows: Bath AS Disease Activity Index (BASDAI) score ≥ 4 and a spinal pain score (BASDAI question 2) ≥ 4 (see Annex 6 for scoring criteria);
5. Subjects who have been treated with non-steroidal anti-inflammatory drugs (NSAIDs) and still have active disease, or who have discontinued NSAIDs due to intolerance; defined as follows: subjects must have had at least 2 cumulative inadequate clinical responses to the recommended dose (≥2 weeks of each NSAID and ≥4 weeks of total use) or intolerance to at least 2 different oral NSAIDs. Intolerance defined as discontinuation of treatment with NSAIDs due to associated adverse events (e.g., allergic reactions, gastrointestinal signs or symptoms, etc.);
6. Subjects taking treatment with NASIDs at the time of screening, requiring stable dose continuation for ≥ 2 weeks prior to randomization; no change in drug dose during the study period except for emergencies; if not taking, discontinuation for at least ≥ 2 weeks prior to randomization;
7. If subjects are enrolled in the study on a combination of methotrexate (MTX), salazosulfapyridine (SASP) and/or hydroxychloroquine (HCQ), subjects must receive a stable dose of MTX (≤25 mg/week) and/or SASP (≤3 g/day) and/or HCQ (≤400 mg/day) for at least 28 days prior to the baseline visit. A maximum of two background csDMARDs allowed in combination;
8. Subjects taking oral glucocorticoids at screening at doses ≤10 mg/day of prednisone (or equivalent doses of other glucocorticoids) that need to be continued for ≥4 weeks prior to randomization; if subjects are not taking oral glucocorticoids, they need to be off them for at least ≥4 weeks prior to randomization;
9. The subject has received ≤ 1 prior treatment with a biologic agent prior to randomization. Subjects previously treated with biologic agents must have been off ≥ 6 half-lives prior to randomization.

Exclusion Criteria:

1. Presence of the following diseases or history of disease:

1. A known or suspected history of complete spinal ankylosis, or clinically and imaging confirmed complete spinal ankylosis;
2. A history of any other autoimmune rheumatic disease;
3. Patients with a combination of severe extra-articular manifestations, such as hyperthermia, interstitial pneumonia, pleurisy, pericarditis, severe vasculitis, or neurological pathology;
4. Patients with current or recent serious, or progressive, or uncontrolled disease, including: hepatic, renal, hematologic, gastrointestinal, endocrine, metabolic, respiratory, cardiovascular, or neurologic disease; or patients who, in the opinion of the investigator, may affect patient safety or compliance;etc.

2.Any of the following laboratory test indicators are met at the time of the screening test:

1. Those who test positive for the following bacteria or viruses at screening, such as HIV, syphilis, Hepatitis B Virus (HBSAg, HBeAg, Hepatitis B Virus-DNA, anyone positive for any of the three), Hepatitis C Virus (positive for anti-Hepatitis C Virus antibodies); If screening stage hepatitis B surface antigen negative (HBsAg-) and anti-hepatitis B core antibody positive (HBcAb+), additional quantitative Hepatitis B Virus-DNA test is required and excluded if quantitative > normal value;
2. Routine blood count: white blood cell count (WBC) <3×109/L, absolute neutrophil count (ANC) <1.5×109/L, absolute lymphocyte count (ALC) <0.8×109/L, platelets (PLT) <100×109/L, hemoglobin (Hb) <100 g/L;etc.

3. Is taking or has a history of taking medication that:

1. Those who are receiving any other csDMARDs or biologic DMARDs (except MTX, SASP, HCQ in the inclusion criteria) or other prohibited concomitant medications; if previous use of csDMARDs such as thalidomide, hydroxychloroquine or leflunomide, those who discontinued thalidomide, hydroxychloroquine, etc. for ≤ 4 weeks and leflunomide for ≤ 8 weeks prior to randomization (using criteria subjects not more than 28 days after Kauleenamine treatment or active carbon elution were not allowed to be enrolled in the trial);
2. Those who have been treated with any tyrosine kinase (JAK) inhibitor (e.g. Tofacitinib, Baricitinib, Upadacitinib, etc.);etc.

4. Those who may be allergic to VC005, similar drugs or their excipients 5. Those with substance abuse or alcohol dependence 6. Subjects who, in the opinion of the investigator, may be at risk of gastrointestinal perforation during the course of the trial 7. Those who have participated in a clinical trial with any drug or device within 12 weeks prior to screening and have used that drug or device 8. Subjects who have a history of major surgery, joint surgery within 6 months prior to screening or who are scheduled to have surgery during the trial 9. Female patients who are planning to become pregnant or who are pregnant or breastfeeding, or who are unable to use effective contraception throughout the trial and for 3 months after the end of the trial (see Appendix 14 for details) 10. Those who, for any reason, are considered by the investigator to be unsuitable for participation in this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2023-04-26 (Actual); Primary Completion 2024-05-11 (Actual); Study Completion 2024-05-11 (Actual)

PRIMARY OUTCOMES:
Percentage of patients achieving ASAS20 | Week 12
  Percentage of patients achieving an Assessment of disease activity (signs and symptoms) in ankylosing spondylitis 20% improvement (ASAS20) in response at week 12 of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Zhanguo Li, Principal Investigator — Peking University People's Hospital; Xu Liu, Principal Investigator — Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China